CLINICAL TRIAL: NCT02523976
Title: Dasatinib Plus Multi-agent Chemotherapy for New Diagnosed Philadelphia Chromosome-positive Acute Lymphoblastic Leukemia
Brief Title: Dasatinib Combined With Chemotherapy in Philadelphia Chromosome-positive Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2015001
Record Dates: First submitted 2015-08-05; First posted 2015-08-14 (Estimated); Last update posted 2026-02-11 (Actual); Status verified 2022-08

CONDITIONS: Acute,Leukemia, Lymphoid
Keywords: Acute; Leukemia; Lymphoid; Philadelphia chromosome; dasatinib
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Philadelphia Chromosome | interventions — Dasatinib; Prednisone; Cyclophosphamide; Daunorubicin; Vincristine; Cytarabine; Mercaptopurine; Methotrexate; Dexamethasone; Mitoxantrone; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): Dasatinib 100 mg per day will be given orally along with combination chemotherapy starting day 8 of induction chemotherapy. Dasatinib will be given continuously (if it's tolerable) for 2 years since achievement of complete remission (CR) as part of consolidation chemotherapy and maintenance therapy.Patients can receive allogeneic hematopoietic stem cell transplantation (HSCT),or patients who keep BCR/ABL negative can receive autologous HSCT whenever possible during their first CR. Otherwise, they will finish the consolidation chemotherapy.
  Interventions: Drug: Dasatinib; Drug: prednisone; Drug: cyclophosphamide; Drug: daunorubicin; Drug: vincristine; Drug: cytarabine; Drug: mercaptopurine; Drug: methotrexate; Drug: dexamethasone; Drug: mitoxantrone; Drug: etoposide; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: autologous hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: Dasatinib — Second-generation tyrosine kinase inhibitor
Drug: prednisone
Drug: cyclophosphamide
Drug: daunorubicin
Drug: vincristine
Drug: cytarabine
Drug: mercaptopurine
Drug: methotrexate
Drug: dexamethasone
Drug: mitoxantrone
Drug: etoposide
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: autologous hematopoietic stem cell transplantation

SUMMARY:
In this single-center, open-label, no control,prospective clinical trial, a total of 30 Philadelphia chromosome-positive acute lymphoblastic leukemia (Ph+ALL) patients will be enrolled. Dasatinib 100 mg per day will be given orally along with combination chemotherapy starting day 8 of induction chemotherapy. Dasatinib will be given continuously (if it's tolerable) for 2 years since achievement of complete remission (CR) as part of consolidation chemotherapy and maintenance therapy.Patients can receive allogeneic hematopoietic stem cell transplantation (HSCT) or autologous HSCT whenever possible during their first CR. Otherwise, they will finish the consolidation chemotherapy. The purpose of current study is to determine the clinical efficacy and tolerability of combination therapy of Dasatinib with multi-agent chemotherapy in newly-diagnosed Ph+ ALL.

DETAILED DESCRIPTION:
In this single-center, open-label, Phase II study, nonrandomized,no control,prospective clinical trial,a total of 30 Philadelphia chromosome-positive acute lymphoblastic leukemia (Ph+ALL) patients will be enrolled.Patients will be diagnosed according to morphologic,immunologic, cytogenetic and molecular(MICM) criteria, including bone marrow morphology, immunophenotype, cytogenetic and molecular genetic (BCR/ABL gene, qualitative and quantitative analysis) examination.

Dasatinib 100 mg per day will be given orally along with combination chemotherapy starting day 8 of induction chemotherapy. Dasatinib will be given continuously (if it's tolerable) for 2 years since achievement of complete remission (CR) as part of consolidation chemotherapy and maintenance therapy.Patients can receive allogeneic hematopoietic stem cell transplantation (HSCT),or patients who keep BCR/ABL negative can receive autologous HSCT whenever possible during their first CR. Otherwise, they will finish the consolidation chemotherapy. Total duration of follow-up will be 2 year after last enrollment.

Pre-treatment evaluation will include complete blood count (CBC) with reticulocyte count, chemistry, electrolytes, coagulation, hepatitis profile, chest X-ray.Evaluation during treatment will include: CBC every two days during myelosuppression, chemistry, electrolytes, coagulation before each cycles of chemotherapy. Quantitative PCR (RQ-PCR) for Bcr-Abl will be done from bone marrow mononuclear cells at diagnosis, at CR, and before each cycles of consolidation chemotherapy,then every 3 months during maintenance therapy. For patients who undergo allogeneic HSCT, quantitative PCR for Bcr-Abl will be done from bone marrow mononuclear cells at the initiation of conditioning, and then every 3 months. PCR will be done in IS standardized lab.

Side effects of combination therapy will be monitored and described according to Common Toxicity Criteria, version 4.0 (National Cancer Institute, USA).

The purpose of current study is to determine the clinical efficacy and tolerability of combination therapy of Dasatinib with multi-agent chemotherapy in newly-diagnosed Ph+ ALL.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 60 years with De novo Philadelphia chromosome positive (Philadelphia chromosome positive or BCR/ABL transcript positive) acute lymphoblastic leukemia.
2. Eastern Cooperative Oncology Group (ECOG) Performance status 2.
3. Adequate end organ function as defined by: Total bilirubin ≤ 1.5 x upper limit of normal（ULN）; serum glutamic-oxaloacetic transaminase(SGOT) and serum glutamic pyruvic transaminase(SGPT) ≤ 2.5 x ULN; Creatinine ≤ 1.5 x ULN; Serum amylase and lipase ≤ 1.5 x ULN; Alkaline phosphatase ≤ 2.5 x ULN unless considered tumor related; Patients must have adequate cardiac function (ejection fraction ≥ 45 % on Multiple Gated Acquisition (MUGA) scan).
4. Patients must have the following laboratory values (≥ lower limit of normal (LLN) or corrected to within normal limits with supplements prior to the first dose of study medication.): Potassium ≥ LLN; Magnesium ≥ LLN; Phosphorus ≥ LLN
5. Patients should sign informed consent form.

Exclusion Criteria:

1. Impaired cardiac function:

   Long QT syndrome or a known family history of long QT syndrome; clinically significant resting brachycardia (<50 beats per minute); ejection fraction < 45 % on MUGA scan. QTc interval > 450 msec on baseline ECG (using the QTcF formula). If QTcF interval>450 msec and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc. Myocardial infarction within 12 months prior to starting study; other clinically significant heart disease (e.g. unstable angina, congestive heart failure or uncontrolled hypertension, uncontrolled arrhythmias).

   Patients who are currently receiving treatment with any medications that have the potential to prolong the QT interval and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug.
2. Other concurrent severe and/or uncontrolled medical conditions:

   Patients with another primary malignant disease, except those that do not currently require treatment; acute or chronic liver, pancreatic or severe renal disease; another severe and/or life-threatening medical disease.
3. Patients who are: (a) pregnant, (b) breast feeding, (c) of childbearing potential without a negative pregnancy test prior to baseline and (d) male or female of childbearing potential unwilling to use contraceptive precautions throughout the trial (post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential).
4. Who is known human deficiency virus (HIV) positive.
5. Use of any other investigational agent in the last 30 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08-01; Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | From date of diagnosis until the date of death from any cause, assessed up to 60 months.

SECONDARY OUTCOMES:
Disease-free survival (DFS) | From the date of complete remission(CR) until the date of documented relapse,assessed up to 60 months.
The complete remission (CR) rate | Participants will be followed for the duration of the treatment, an expected average of 6 months.
The molecular CR rate | Participants will be followed for the duration of the treatment, an expected average of 24 months.
The plasma level of dasatinib in the regimen | Up to 3 months.
The Cerebrospinal fluid level of dasatinib in the regimen | Up to 6 months.
Number of adverse event of combined treatment | Participants will be followed for the duration of the treatment, an expected average of 24 months.
Grade of adverse event of combined treatment | Participants will be followed for the duration of the treatment, an expected average of 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Dr., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Gong X, Li L, Wei H, Liu B, Zhou C, Zhang G, Liu K, Lin D, Gong B, Wei S, Li Y, Mi Y, Wang Y, Wang J. A Higher Dose of Dasatinib May Increase the Possibility of Crossing the Blood-brain Barrier in the Treatment of Patients With Philadelphia Chromosome-positive Acute Lymphoblastic Leukemia. Clin Ther. 2021 Jul;43(7):1265-1271.e1. doi: 10.1016/j.clinthera.2021.05.009. Epub 2021 Jun 10. PMID 34120773
- [Derived] Zhang GJ, Gong XY, Qiu SW, Zhou CL, Liu KQ, Lin D, Liu BC, Wei H, Wei SN, Li Y, Gu RX, Gong BF, Liu YT, Fang QY, Mi YC, Wang Y, Wang JX. [Dasatinib combined with multi-agent chemotherapy regimen in newly diagnosed Philadelphia chromosome-positive acute lymphoblastic leukemia: a prospective study from a single center]. Zhonghua Xue Ye Xue Za Zhi. 2021 Feb 14;42(2):109-115. doi: 10.3760/cma.j.issn.0253-2727.2021.02.004. Chinese. PMID 33858040